CLINICAL TRIAL: NCT04804475
Title: Effects of Square-stepping Exercise Training on the Attention, Dynamic Balance and Lower Extremity Motor Coordination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Gulsum Tikac, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Effect of SSE Training
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2021-03

CONDITIONS: Sedentary Healthy Young Individuals
Keywords: Square-stepping exercise training; attention; dynamic balance; motor coordination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Active Comparator): Throughout 3 weeks SSE training was administered 4 days a week for a length of 45 minutes in each session. All the analyses were conducted at the start and at the end of 3-week long training.
  Interventions: Other: Exercise Trainig
- Control Group (No Intervention): This group has no intervention. Evaluations were only made at the start and at the end of 3-week long.

INTERVENTIONS:
Other: Exercise Trainig — SSE is performed on a thin exercise mat divided into 40 small squares in 250 cm x 100 cm of size (25 cm each part). Participants are given patterns of a few steps and asked to take steps that match them. Participants must, in principal, move ahead in line with the length forward with no contact on the lines forming the squares. Forward, backward, lateral and oblique stepping patterns are required. Stepping patterns get increasingly difficult. Each pattern consists of 2 to 16 steps; participants are asked to repeat step pattern till the end of exercise mat. Upon completing a pattern, another pattern in the same mirror-image is repeated. In essence each pattern is reiterated for 3-5 times and next its mirror-image pattern is repeated but if participants face challenge in performing the pattern it is repeated till the pattern is learnt
  Other Names: Square-steeping exercise
  Arms: Training Group

SUMMARY:
Physical activity plays an indispensable role to lead a healthy life. Square-stepping exercises (SSE) are aerobic exercises. Our study was designed to investigate the effects of square-stepping exercise training on the attention, dynamic balance and lower extremity motor coordination of sedentary healthy young individuals.

A total of 112 volunteers within the age range of 20-25 participated in the research. Participants were randomly divided into two groups, as 56 participants were study group (28 females, 28 males) and 56 participants were control group (28 females, 28 males). Demographic data and exercise habit of the individuals were documented. Stroop Test was used to assess Attention, Four-step Square Test was used to assess Dynamic Balance and Lower-extremity Motor Coordination Test was used to assess Motor Coordination. Throughout 3 weeks SSE training was administered 4 days a week for a length of 45 minutes in each session. All the analyses were conducted at the start and at the end of 3-week long training.

DETAILED DESCRIPTION:
Demographic data and exercise habit of the individuals were documented. Stroop Test: The Stroop test measures cognitive functions such as cognitive flexibility, attention, inhibition, and reaction time. The test is administered by asking participants to name the colors of words written in different colors; they must focus on the colors of the words, not their meanings. Research has shown that age significantly affects processing speed and reaction time, especially in children aged 5-15 and adults aged 20-82.

Four-step Square Test: The subject is required to sequentially step over four canes set-up in a cross configuration on the ground. At the start of the test, the subject stands in Square 1 facing Square 2. The aim is to step as fast as possible into each square with both feet in the following sequence: Square 2, 3, 4, 1, 4, 3, 2, 1 (clockwise to counterclockwise).

Lower-extremity Motor Coordination Test was developed as an easy, yet effective tool to clinically assess, measure, and evaluate the deficits in Lower Limb Motor Coordination

ELIGIBILITY:
Inclusion Criteria:

* Being within the age range of 20-25,
* Not continuing any exercise program for the last 1 year,
* Not having any disease impacting neurological, orthopedic or lower extremity system,
* Not having surgery history on lower extremity,
* Not having visual and hearing problem.

Exclusion Criteria:

* Having visual and hearing problem,
* Neurological problem debilitating one's walking,
* Having psychiatric or orthopedic problem
* Having surgery history on lower extremity.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Attention Assessment (Stroop test) | 3 weeks
  The Stroop test measures cognitive functions such as cognitive flexibility, attention, inhibition, and reaction time. The test is administered by asking participants to name the colors of words written in different colors; they must focus on the colors of the words, not their meanings.
Dynamic Balance Assessment (Four-step Square Test) | 3 weeks
  The subject is required to sequentially step over four canes set-up in a cross configuration on the ground.
  At the start of the test, the subject stands in Square 1 facing Square 2. The aim is to step as fast as possible into each square with both feet in the following sequence: Square 2, 3, 4, 1, 4, 3, 2, 1 (clockwise to counterclockwise)
Motor Coordination Assessment (Lower extremity Motor Coordination Test) | 3 weeks
  This test is completed with the patient sitting.There are two red targets on a sheet, 6 cm in diameter each, which are placed 30 apart in a vertical direction. The patient, sitting in a comfortable position with their knees flexed at 90 degrees and their heels on the proximal target, is asked to alternately move their leg back and forth to accurately touch the red target with their big toe. They must do this as quick as they can, and as many times as they can, in 20 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Gulsum Tikac, Principal Investigator — Pamukkale University; Ayse Unal, Study Director — Pamukkale University; Filiz Altug, Study Chair — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tikac G, Unal A, Altug F. Effects of Square-Stepping Exercise Training on the Attention, Dynamic Balance and Lower Extremity Motor Coordination. Physiother Res Int. 2026 Jan;31(1):e70123. doi: 10.1002/pri.70123. PMID 41216663